CLINICAL TRIAL: NCT03175965
Title: Characteristics of the Somatosensory Evoked Potentials Indicating Poor Neurologic Outcome After Cardiac Arrest
Brief Title: Prognostic Value of P30 After Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Uijeongbu St. Mary Hospital (Other)
Collaborators: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Joo Suk Oh, MD. PhD., Associate Professor, Uijeongbu St. Mary Hospital
Other Study IDs: XC17OEDI0009
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Heart arrest, hypothermia, SEP, prognosis
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Somatosensory evoked potential — Somatosensory evoked potential on 24, 72 hours after cardiac arrest.

SUMMARY:
This study aims to examine whether P30 wave of somatosensory evoked potentials (SEP) is related with outcome after cardiac arrest. The study design is a prospective, multicenter-observational study. Patients survived after out-of-hospital cardiac arrest undergoing hypothermic-targeted temperature management will participate in the study. Relationship of P30 wave of SEP with the neurologic outcome on hospital discharge will be evaluated.

DETAILED DESCRIPTION:
The absence of N20 of the somatosensory evoked potentials (SEP) is recommended as a valuable predictor of poor neurologic outcome in post-cardiac arrest patients. However, interpretation of N20 is affected by the background noise levels. Reliable analysis of N20 is limited with high noise levels and artifacts. Moreover, presence of N20 does not guarantee good neurologic outcome. P30 is a positive deflection of N20 occurring on 25-35 msec. According to our pilot study, N20 without following P30 is related with poor outcome, while N20 followed by P30 is highly related with good outcome. P30 is evident even when the N20 is ambiguous in patients with good outcome. We hypothesized that the negative-positive deflection of N20-P30 components is more valuable predictor than the N20 alone. In this observational study, we will identify whether presence of P30 checked on 24 and 72 hours after cardiac arrest predicts neurologic outcome more accurately than the presence of N20 alone.

ELIGIBILITY:
Inclusion Criteria:

* Comatose survivors after out-of-hospital cardiac arrest

Exclusion Criteria:

* Not treated by hypothermic-targeted temperature management

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out-of-hospital cardiac arrest patients undergoing hypothermic-targeted temperature management in the four academically affiliated tertiary care centers .
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Association of abscence of P30 with poor outcome without under the influence of hypothermia and sedation | 72 hours after ROSC
  SEP under the normothermic-TTM without sedation

SECONDARY OUTCOMES:
Association of abscence of P30 with poor outcome under the influence of hypothermia and sedation | 24 hours after ROSC
  SEP under the hypothermic-TTM with sedation
Association of N20 with high amplitude with poor outcome without under the influence of hypothermia and sedation | 72 hours after ROSC
  SEP under the normothermic-TTM without sedation
Association of N20 with high amplitude with poor outcome under the influence of hypothermia and sedation | 24 hours after ROSC
  SEP under the hypothermic-TTM with sedation

CONTACTS AND LOCATIONS:
Overall Officials: Joo Suk Oh, MD, Study Chair — Uijeongbu St. Mary's Hospital
Locations (4):
- South Korea (4):
  - Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si, Gyeonggi-do
  - Seoul St. Mary's Hospital, Seoul
  - Yeouido St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No